CLINICAL TRIAL: NCT05310279
Title: Feasibility of An Active Video Gaming Intervention to Improve Health and Function in Adults With Mobility Impairments
Brief Title: Feasibility of An Active Video Gaming Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Researcher, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300009049; 90REGE000 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Physical Disability
Keywords: Exergaming, Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active video gaming (Experimental): Participants will engage in 6 weeks of active video gaming (AVG), 2x/week
  Interventions: Other: GAIMplank

INTERVENTIONS:
Other: GAIMplank — The GAIMplank video game controller will be used to play active video games.

SUMMARY:
Replacing sedentary behaviors during leisure time with active video gaming (AVG) has been shown to be an enjoyable option for increasing the amount of physical activity acquired each week. This project will examine the feasibility of an AVG intervention using the GAIMplank.

DETAILED DESCRIPTION:
Replacing sedentary behaviors during leisure time with active video gaming (AVG) has been shown to be an enjoyable option for increasing the amount of physical activity acquired each week. A growing body of literature indicates that increases in energy expenditure can be achieved during AVG play in people with physical disabilities, including those with mobility impairments such as cerebral palsy (CP), spinal cord injury, stroke, and other neurological conditions. AVGs are particularly important for people with disabilities given the higher rate of inaccessible features in the built environment and the difficulty in finding activities they enjoy. Since AVG devices are relatively affordable, they also hold promise as a scalable product for promoting higher levels of physical activity and fitness among people with disabilities.

There continues to be a pressing need to make gaming controllers accessible to people who are unable to stand for long periods, cannot stand on a small platform due to poor balance or extreme obesity, or who are unable to stand and are full-time wheelchair users. The GAIMplank controller, was developed and tested for usability among people with mobility impairments. During usability testing, a sample of 21 adults were able to successfully access and play a series of standard PC video games using trunk/body movements to produce game play action. Using validated survey tools, participant usability scores and qualitative feedback indicated above average usability for the GAIMplank system. In addition, participants enjoyed the activity and reported game play as light to moderate intensity activity.

This project will examine the feasibility of an AVG intervention using the GAIMplank.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Self-reported physical disability that limits their mobility
* Communicate in English

Exclusion Criteria:

* Significant impairment in visual acuity that prevents seeing a 52" TV screen to follow exercise
* Body weight >400 lbs
* Cognitive or linguistic problems with understanding instructions or filling in self-administered outcome measures in English as determined by a score of <17 on the telephone-version of the Mini-Mental State Exam
* Any other conditions that would limit ability to play video games
* Cardiovascular disease event within the past 6 months
* Severe pulmonary disease or renal failure
* Currently pregnant
* Ongoing exacerbation of a health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Level of physical activity from baseline to 6 weeks | 6 weeks
  Instrument physical activity questionnaire - disability (IPAQ-D)

SECONDARY OUTCOMES:
Physical activity enjoyment from baseline to 6 weeks | 6 weeks
  Physical activity enjoyment scale
Health-related quality of life from baseline to 6 weeks | 6 weeks
  SF-36v2

CONTACTS AND LOCATIONS:
Locations (1):
- WHARF, Homewood, Alabama, United States

IPD SHARING:
Plan to Share IPD: No